CLINICAL TRIAL: NCT05006092
Title: Multicenter Evaluation Study of the CADe System ENDOMIND in Surveillance Endoscopy for Colorectal Cancer in German Outpatient Cohort
Brief Title: Surveillance Modified by Artificial Intelligence in Endoscopy (SMARTIE)
Acronym: SMARTIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Klinikum Stuttgart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: F-2021-047
Record Dates: First submitted 2021-06-11; First posted 2021-08-16 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Surveillance Endoscopy for Colorectal Cancer; Artificial Intelligence; Polyps of Colon; CADe
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surveillance endoscopy with CADe support (Experimental): Endoscopy perfomed with CADe support.
  Interventions: Device: ENDOMIND
- conventional surveillance endoscopy (No Intervention): Endoscopy perfomed without CADe support.

INTERVENTIONS:
Device: ENDOMIND — CADe system for Polyp detection
  Arms: surveillance endoscopy with CADe support

SUMMARY:
Evaluation of an artificial intelligence system for polyp detection (CADe)

DETAILED DESCRIPTION:
We aim to evaluate the artificial intelligence system ENDOMIND that supports endoscopist in detection of polyps during surveillance endoscopy for colorectal cancer. 1070 patients out of 6 gastroenterologic practice are randomized 1:1 for conventional surveillance colonoscopy vs. surveillance with AI support. Primary endpoint is Adenoma detection rate.

ELIGIBILITY:
Inclusion Criteria:

* indication CRC surveillance endoscopy
* indication post-polypectomy surveillance endoscopy
* positive fecal immunochemical test in patients >=50 years

Exclusion Criteria:

* reasonable suspicion of inflammatory bowl disease
* reasonable suspicion of familiar polyposis Syndrome
* Patient after radiation/resection of colonic parts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1149 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | 4 months
  proportion of individuals undergoing a complete screening colonoscopy who have one or more adenomas

SECONDARY OUTCOMES:
polyp detection rate | 4 months
  Exmainations with minimum one polyp detected.
withdrawal time | 4 months
  Time of withdrawal.
resection time | 4 months
  Time spent on polyp resections.
Boston Bowl Preparation Score | 4 months
  minimum 0, Maximum 9; should be higher than 5 for appropriate surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hann, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Universitätsklinikum Würzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lux TJ, Banck M, Sassmannshausen Z, Troya J, Krenzer A, Fitting D, Sudarevic B, Zoller WG, Puppe F, Meining A, Hann A. Pilot study of a new freely available computer-aided polyp detection system in clinical practice. Int J Colorectal Dis. 2022 Jun;37(6):1349-1354. doi: 10.1007/s00384-022-04178-8. Epub 2022 May 11. PMID 35543874